CLINICAL TRIAL: NCT02905448
Title: Effects of an ad Libitum Consumed Low-fat Plant-based Diet Supplemented With Plant-based Meal Replacements on Variety of Risk Factors for Chronic Non-communicable Diseases
Brief Title: Low Fat Plant-Based Supplemented Diet Effects on Risk Factors for Chronic Non-communicable Diseases
Acronym: LFPBDS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Jakše s.p. (Other)
Responsible Party: Principal Investigator, Boštjan Jakše, PE teacher (PhD student), Barbara Jakše s.p.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KR2
Record Dates: First submitted 2016-09-02; First posted 2016-09-19 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Hyperlipidemia; Metabolic Syndrome X
Keywords: Obesity; Body composition; Atherosclerosis; Insulin resistance; Hyperuricemia
MeSH Terms: conditions — Hyperlipidemias; Metabolic Syndrome; Obesity; Atherosclerosis; Insulin Resistance; Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low fat plant-based diet (Experimental): Low fat plant-based nutrition: low fat plant-based diet supplemented with plant-based meal replacements
  Interventions: Other: Low fat plant-based nutrition

INTERVENTIONS:
Other: Low fat plant-based nutrition — Conventional low fat plant-based meals free from animal source foods three times daily.
  Plant-based meal replacement with Herbalife European Free From Vanilla formula two times daily.
  Herbal beverage two times daily. Dietary fiber supplements is taken three times daily (10-36w) and more high fat whole plant-based foods (avocado, tofu, seeds) Conventional food intake is taken ad libitum and no calorie counts or restrictions will be applied.
  From 10 to 36 weeks we added vitamin B12 and EPA+DHA fatty acid
  Other Names: LFPBD

SUMMARY:
The effect of a diet free from animal-sourced nutrients on a variety of risk factors for chronic non-communicable diseases in weight reduction programs is not well established. In this non-randomised interventional study, the investigators will document the effects of a low-fat, plant-based diet supplemented with two daily plant-based meal replacements on serum LDL cholesterol as a primary end-point and total cholesterol, triglycerides, serum fasting glucose, serum urate, serum insulin-like growth factor 1 (IGF-1) and body fat mass as secondary end-points. These end-points will be measured at baseline, after 10 weeks and after 36 weeks of intervention. Participants will be enrolled in the interventional arm with prescribed low fat plant-based diet from the group of all applicants to a free living population-based diet optimising program. The choice to participate in the study will be made by participants themselves.

The investigators hypothesise that low-fat plant based diet supplemented with plant-based meal replacements eaten ad libitum allows a significant reduction of serum LDL cholesterol concentration.

DETAILED DESCRIPTION:
This study is designed as a non-randomized, interventional 36 week trial. The dietary intervention is executed in free living conditions with participants engaging in their regular daily work and social activities.

The dietary intervention was executed in free-living conditions with participants engaging in their regular daily work and social activities. The plant-based dietary plan included 2 plant-based meal replacement and 3 conventional meals based on starch nutrients (potatoes, sweet potatoes, rice, oatmeal, whole-grain pasta, beans, peas, lentils, and similar ones), fruits (seasonal fruits and various berries), and nonstarch vegetables (color and leafy vegetables). Spices and tomato sauce (without oil) and one regular-sized spoon of flaxseed were recommended as well. The participants were recommended to consume no more than 5-6 grams of salt per day. All milk and dairy products, vegetable oils, and fats were excluded from the diet. Meat was allowed (but not recommended) once weekly to relieve social pressures on participants which they often encountered from their circle of influence (i.e., family, friends, and coworkers) when changing the diet to plant-based sources. The total macronutrient composition of the intervention diet was approximated to 15% protein, 70% carbohydrates, and 15% fat. No soybean was included in first 10 weeks of intervention. Dietary fiber content was approximated to 40-45 g per day. Both meal replacements and conventional meals were allowed to be consumed ad libitum (to full satiety). No calorie count or limits were instituted. Additionally, two herbal drinks daily containing black, green and hibiscus tea extracts were added to the intervention.

After 10 weeks, we have added to the interventional diet EPA and DHA omega 3 fatty acids (once per day 3 tbl or 567 mg per 1 tbl), vitamin B12 - methylcobalamin (1000 mcg twice a week) and additional intake of dietary fiber supplement powder (three times a day of 5 g) on supplement side and a larger selection of moderate amount of high fat whole plant-based foods (e.g. avocado, soybean tofu, sesame seeds, almonds) at the conventional side.

No calorie count or limits are instituted to test the hypothesis that ad libitum intake of interventional diet allows significant body fat reduction and improvement variety of risk factors for chronic non-communicable diseases.

All participants will be followed at weekly intervals for body composition indices and at 10 and 36 weeks for serum biochemical end-points.

Evaluation of dietary diaries and meal photographs will be used to correct and adjust deviations from the targeted dietary plan and to help participants prepare the meals according to the dietary plan.

ELIGIBILITY:
Inclusion Criteria:

* Self selected free living participants older than 18 years of age
* Non overweight, overweight, obese
* Sign informed consent for participation in the study

Exclusion Criteria:

* Pregnant or lactating women, patients with dietary restrictions from a treating physician and patients with active malignant disease were excluded from the study
* Already on plant-based (vegan) diet
* Competitive or top level athletes
* Subjects already taking part in any other interventional dietary program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Serum LDL cholesterol concentration change from baseline | Baseline, 10 weeks and 36 weeks

SECONDARY OUTCOMES:
Serum total cholesterol concentration change from baseline | Baseline, 10 weeks and 36 weeks
Serum triglyceride concentration change from baseline | Baseline, 10 weeks and 36 weeks
Fasting serum glucose concentration change from baseline | Baseline, 10 weeks and 36 weeks
Serum uric acid concentration change from baseline | Baseline, 10 weeks and 36 weeks
Serum IGF-1 concentration change from baseline | Baseline, 10 weeks and 36 weeks
Body fat mass change from baseline | Baseline, 10 weeks and 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bostjan Jakse, PE teacher, Principal Investigator — Barbara Jakse s.p.

IPD SHARING:
Plan to Share IPD: Yes
Data will be open to public if demanded by the publication/journal.

REFERENCES:
- [Background] Wang F, Zheng J, Yang B, Jiang J, Fu Y, Li D. Effects of Vegetarian Diets on Blood Lipids: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2015 Oct 27;4(10):e002408. doi: 10.1161/JAHA.115.002408. PMID 26508743
- [Background] Li Z, Treyzon L, Chen S, Yan E, Thames G, Carpenter CL. Protein-enriched meal replacements do not adversely affect liver, kidney or bone density: an outpatient randomized controlled trial. Nutr J. 2010 Dec 31;9:72. doi: 10.1186/1475-2891-9-72. PMID 21194471
- [Background] Jakse B, Jakse B, Pajek J, Pajek M. Effects of ad libitum consumed, low-fat, high-fiber plant-based diet supplemented with plant-based meal replacements on cardiovascular risk factors. Food Nutr Res. 2019 May 21;63. doi: 10.29219/fnr.v63.1560. eCollection 2019. PMID 31191190